CLINICAL TRIAL: NCT03613584
Title: A Double-blind, Placebo-controlled Pilot Trial to Investigate the Administration of Von Willebrand Factor Concentrate (Willfact®, LFB France) in Adult Patients During Extracorporeal Membrane Oxygenation
Brief Title: Von Willebrand Factor Concentrate During ECMO Support
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tirol Kiniken GmbH (Other)
Collaborators: LFB BIOMEDICAMENTS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ECMO-vWFC
Record Dates: First submitted 2018-03-22; First posted 2018-08-03 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Acquired Von Willebrand Disease
MeSH Terms: interventions — von Willebrand Factor; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The vWFC or placebo will be prepared by the local hospital pharmacy or independent nurses from another ward (on holidays and weekends). To keep the blinding for the treating physicians and the study team syringes and lines with light protection (orange color) will be used. So the color of the medication (colorless to slightly yellowish) cannot be distinguished.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group W (von Willebrand factor concentrate) (Active Comparator): The patient receives von Willebrand factor concentrate (vWFC) as a bolus of 25 IU/kg followed by a continuous infusion of 50 IU/kg/24h until the weaning from ECMO is completed or if ECMO is needed longer than 7 days, the administration of the Investigational Medicinal Product (IMP) will be stopped on the 7th day.
  Interventions: Drug: Von Willebrand Factor
- Group S (standard therapy with saline solution) (Placebo Comparator): The patient receives the standard therapy plus an additional volume of saline solution equivalent to the amount of von Willebrand factor concentrate (vWFC) the patient would receive in Group W to keep the blind. The volume is given according to the VWFC-solution (0.25 ml/kg BW) what would be resulting from the patient's weight followed by a continuous saline infusion (0.50 ml/kg BW) until the weaning from ECMO is completed or if ECMO is needed longer than 7 days, the Investigational Medicinal Product (IMP) administration is stopped on the 7th day.
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: Von Willebrand Factor — Bolus and continuous infusion of the Investigational Medicinal Product (IMP) during extracorporeal membrane oxygenation (ECMO)
  Arms: Group W (von Willebrand factor concentrate)
Drug: Saline Solution — Bolus and continuous infusion of the Investigational Medicinal Product (IMP) during extracorporeal membrane oxygenation (ECMO)
  Arms: Group S (standard therapy with saline solution)

SUMMARY:
During treatments with extracorporeal circuits such as extracorporeal membrane oxygenation (ECMO) degradation of high molecular weight (HMW) of von Willebrand factor (vWF) multimers occur leading to an acquired von Willebrand disease. This disease is associated with increased bleeding and requirement for the transfusion with allogenic blood products especially packed red blood cells (PRBCs). A continuous treatment with von Willebrand factor concentrate (vWFC) may restore the multimers and bleeding can be avoided. Therefore a randomized, double-blind, prospective, controlled, two-arm clinical trial was designed, comparing patients receiving vWFC versus placebo.

DETAILED DESCRIPTION:
Increased shear stress during mechanical circulatory support (MCS) by extracorporeal membrane oxygenation (ECMO) and ventricular assist devices (VAD) can provoke premature degradation of high molecular weight (HMW) of von Willebrand factor (vWF) multimers. In patients with intractable cardiac and/or respiratory failure requiring emergency ECMO support, the investigators recently demonstrated an essential decrease in high molecular weight (HMW) vWF multimer bands 24 and 48 hours after initiation of ECMO compared to baseline. Blood loss and transfusion requirement during and shortly after ECMO support may be strengthened by loss of HMW vWF multimers.

Administration of vWF concentrates may support restoration of primary hemostasis in patients during ECMO support. Consequently the need for packed red blood cells (PRBCs) during ECMO support may be reduced thus positively influencing morbidity and mortality of ECMO patients. The investigators hypothesize, that treatment with vWF concentrate reduces the need for PRBCs during ECMO support. Therefore the primary aim of this clinical trial is to find out if the need of PRBCs differs in the group receiving a von Willebrand factor concentrate (vWFC), or the placebo group (saline).

This clinical trial is planned as a randomized, double-blind, prospective, controlled, two-arm, two-center study. Patients with intractable cardiac and/or respiratory failure requiring emergency ECMO support undergoing surgery (Department of Anaesthesiology and Intensive Care Medicine) or treated at the General and Surgical Intensive Care Unit (ACI), Traumatologic Intensive Care Unit (TICU), Cardiologic Intensive Care Unit (CCU) or the ICU of the Department of Visceral, Transplant and Thoracic Surgery at the Hospital Innsbruck (Tirol Kliniken GmbH), Austria will be enrolled in the study when meeting the inclusion- and exclusion criteria. If a patient meets the inclusion criteria and is recruited for the study, the patient will be randomized either to the group receiving vWFC or placebo S. Before the implementation of the ECMO the Baseline investigations need to be conducted. As soon as they are completed the ECMO cannula can be inserted.

The administration of the Investigational Medicinal Product (IMP) will be start within 24h after ECMO installation. Directly before IMP-start blood samples (Visit 2) will be drawn. After 24h (Visit 3), 60h (Visit 4) and on day 5 (Visit 5) of the start of the study medication visits will be conducted, whereas on day 5 (Visit 5) no special laboratory (measurement of HMW vWF) will be analyzed. If ECMO can be terminated, a visit (Visit 6) directly before the stop of the ECMO will be conducted. 36 h after the termination of the ECMO Visit 7 (termination) will be performed. If the ECMO is needed longer than 7 days, the administration of the IMP will be stopped on day 7 and a visit after 36 hours of IMP-stop will be done for safety reasons but without special laboratory. After 30 days an interview will be performed with the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the need of veno-arterial or veno-venous ECMO for a minimum of 48 hours
* Age ≥ 18 years

Exclusion Criteria:

* Patient with known thromboembolic event in the last 30 days
* Inevitable lethal course
* Severe Liver failure: Quick < 30 %
* Pregnancy
* Patient with known refusal of a participation in this clinical trial
* Active participation in another clinical trial
* Any condition, including the presence of laboratory abnormalities, which would place the subject at unacceptable risk if he/she were to participate in the study or confound the ability to interpret data from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2018-04-16 (Actual); Primary Completion 2021-03-10 (Estimated); Study Completion 2021-03-10 (Estimated)

PRIMARY OUTCOMES:
Transfusion requirement of PRBC | Between start of IMP (Visit 2) until 24 hours after IMP-start (Visit 3)
  Difference in the number of red blood cells concentrates between the treatment arms per day

SECONDARY OUTCOMES:
Transfusion requirements of other allogenic blood products | Between start of ECMO (Visit 1) and 36 hours after ECMO Stop (Visit 7)
  Difference in the number of other high risk allogenic transfusion products (fresh frozen plasma and platelet concentrate) between the treatment arms per day
Requirements of coagulation factor concentrates | Between start of ECMO (Visit 1) and 36 hours after ECMO Stop (Visit 7)
  Amount of coagulation factor concentrates given during ECMO support between the treatment arms per day
Number of vWF-HMW multimer bands | Between start of ECMO (Visit 1) and 36 hours after ECMO Stop (Visit 7)
  Number of vWF multimer bands measured via SDS-agarose gel electrophoresis between the treatment arms
Assessment of thromboelastometry | Between start of ECMO (Visit 1) and 36 hours after ECMO Stop (Visit 7)
  Difference in thromboelastometry between the treatment arms
Changes in thrombocytes | Between start of ECMO (Visit 1) and 36 hours after ECMO Stop (Visit 7)
  Difference in platelet number
Renal function | Between start of ECMO (Visit 1) and 36 hours after ECMO Stop (Visit 7)
  Difference in the daily urine output
Number of participants with bleeding events | Between start of ECMO (Visit 1) and 36 hours after ECMO Stop (Visit 7)
  Number of patients with bleeding events assessed by a bleeding score based on Mazzeffi et al 2013
Assessment vWF-HMW function | Between start of ECMO (Visit 1) and 36 hours after ECMO Stop (Visit 7)
  vWF function (vWF:Ag, vWF:RCo, and F:VIII) via photooptical measurement between the treatment arms
Assessment of activated partial thromboplastin time (aPTT) assay | Between start of ECMO (Visit 1) and 36 hours after ECMO Stop (Visit 7)
  aPTT assay [seconds] between the treatment arms
Changes in red blood cell number | Between start of ECMO (Visit 1) and 36 hours after ECMO Stop (Visit 7)
  Differences in red blood cell number and hemoglobin between the treatment arms
Number of participants with thromboembolic events | 36 hours after IMP-Stop
  Number of participants with thromboembolic events as assessed via duplex ultrasonic investigation of the cervical vessels (Carotis und Vertebralis) and major leg veins
Assessment of Prothrombin time (PT) assay | Between start of ECMO (Visit 1) and 36 hours after ECMO Stop (Visit 7)
  PT assay [%] between the treatment arms
Assessment of activated clotting time (ACT) | Between start of ECMO (Visit 1) and 36 hours after ECMO Stop (Visit 7)
  ACT assay [seconds] between the treatment arms

CONTACTS AND LOCATIONS:
Locations (2):
- Austria (2):
  - Medical University Innsbruck / Department for Anesthesia and Intensive Care Medicine, Innsbruck
  - Medical University Innsbruck / Department for General and Surgical Critical Care Medicine, Innsbruck

REFERENCES:
- [Background] Tauber H, Streif W, Fritz J, Ott H, Weigel G, Loacker L, Heinz A, Velik-Salchner C. Predicting Transfusion Requirements During Extracorporeal Membrane Oxygenation. J Cardiothorac Vasc Anesth. 2016 Jun;30(3):692-701. doi: 10.1053/j.jvca.2016.01.009. Epub 2016 Jan 11. PMID 27321792
- [Background] Tauber H, Ott H, Streif W, Weigel G, Loacker L, Fritz J, Heinz A, Velik-Salchner C. Extracorporeal membrane oxygenation induces short-term loss of high-molecular-weight von Willebrand factor multimers. Anesth Analg. 2015 Apr;120(4):730-6. doi: 10.1213/ANE.0000000000000554. PMID 25565317
- [Background] Velik-Salchner C, Eschertzhuber S, Streif W, Hangler H, Budde U, Fries D. Acquired von Willebrand syndrome in cardiac patients. J Cardiothorac Vasc Anesth. 2008 Oct;22(5):719-24. doi: 10.1053/j.jvca.2007.05.013. Epub 2007 Aug 3. No abstract available. PMID 18922429